CLINICAL TRIAL: NCT01107678
Title: The YMCA After School Program of Physical Activity and Nutrition
Brief Title: YMCA-Physical Activity and Nutrition
Acronym: YMCA-PAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSCL16198; R01DK074909 (NIH)
Record Dates: First submitted 2010-03-26; First posted 2010-04-21 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Childhood Obesity
Keywords: YMCA; Preventative child obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YMCA PAN (Experimental): YMCA PAN (Physical activity and nutrition)- Consists of organized physical activity and controlled serving sizes of healthy low fat snacks
  Interventions: Other: Healthy Snacks and Organized Physical Activity
- YMCA Standard CAre (Experimental): YMCA standard care - Follow the standard care of the YMCA after school Y-Care program for physical activity and nutrition
  Interventions: Other: Healthy Snacks and Organized Physical Activity

INTERVENTIONS:
Other: Healthy Snacks and Organized Physical Activity — Children in the intervention group will receive healthy snacks, smaller portion sizes and participate in organized physical activity on a daily bais
  Other Names: YMCA PAN; YMCA Standard Care

SUMMARY:
There is an epidemic rise in the number of overweight and obese children. Overweight and obesity in children tracks into adulthood and carries elevated risk of chronic diseases such as seen with the metabolic syndrome (i.e., elevated glucose, hypertension, etc.). Low levels of PA and poor nutrition seem to be tightly linked to the increase in overweight and obesity. A minimal intervention that targets simple strategies for both sides of the energy balance equation may diminish overweight and obesity. Increasing moderate to vigorous physical activity and improving nutrition through snacks is a feasible, low cost strategy and can be disseminated nationally through the YMCA, if successful. Specifically, we expect that children receiving YMCA PAN will show smaller changes in BMI after 3 years of the intervention when compared to children not receiving YMCA PAN (i.e. standard, existing YMCA After School Program or "YMCA standard care").

DETAILED DESCRIPTION:
Our primary outcome measurement is body mass index (BMI) as this is now recommended by major health organizations as the preferred measure for the determination of obesity. All children at YMCA After School Programs will receive either YMCA-PAN or YMCA standard care; however, we will only follow children in grades kindergarten through second grade (K-2). For children in grades K-2, we will determine if 3 years of increased physical activity and snacks lower in energy and fat and higher in nutrient density will diminish gains in BMI. We have specifically targeted an increase of moderate to vigorous physical activity (MVPA) by 225 minutes per week that is delivered in YMCA-PAN as this is a compromise between the recommendations suggested by Healthy People 2010 and the Institute of Medicine (IOM) and is administratively feasible within the existing YMCA After School Programs. YMCA-PAN would exceed the Healthy People 2010 guidelines and would provide the majority of PA for the IOM guidelines. Children would satisfy the IOM guidelines with just 15 additional minutes of MVPA accrued throughout the day in physical education class or free play. Finally, YMCA PAN would provide opportunity for PA at the very time the guidelines call "most critical:" the hours between 3 and 6pm when children have finished the school day and frequently are sedentary. For the nutritional component, we are targeting snacks, as snacks are part of the YMCA after school programs, snacks contribute significantly to 24 hour energy intake, children are increasingly in control of the snacks they consume, and we have previously diminished 24 hour energy intake and fat intake using snacks in elementary school children.

We will provide this intervention using regular YMCA staff and use the regular time periods for PA that exist in the YMCA after school programs. We will also use the regular YMCA staff to provide snacks. Specifically, we expect that children receiving YMCA-PAN will show smaller changes in BMI after 3 years of the intervention when compared to children not receiving YMCA-PAN (i.e. standard, existing YMCA after school program or "YMCA standard care").

ELIGIBILITY:
Inclusion Criteria:

* kindergarten through second grade age;

Exclusion Criteria:

* no BMI requirements but must meet age requirements and be available throughout the duration of the study

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 966 (Actual)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 3 years
  Body weight and height will be measured in order to calculate BMI

SECONDARY OUTCOMES:
Daily physical activity levels | Daily
  Length of time and intensity of the program's physical activity sessions will be measured by visual observation on a daily basis
Daily energy intake | Daily
  Energy intake of the snacks served during the program will be measured by visual observation in both the intervention and control schools on a daily basis

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Donnelly, EdD, Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States